CLINICAL TRIAL: NCT00001873
Title: Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation Followed by T-Cell Add-Back for Hematological Malignancies - Role of Cyclosporine
Brief Title: The Role of Cyclosporine in Blood Cell Transplants With T-Cell Add-Back for Blood Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 990046; 99-H-0046
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2017-06-13

CONDITIONS: Chronic Lymphocytic Leukemia; Graft vs Host Disease; Hematologic Neoplasm; Multiple Myeloma; Myelodysplastic Syndrome
Keywords: Peripheral Blood Stem Cells; Cyclosporine; Cyclosphosphamide; Whole Body Irradiation; Donor Apheresis; Leukemic Relapse; Graft vs. Host Disease; Graft-Versus-Leukemia; Graft-Versus-Myeloma; Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndromes; Multiple Myeloma; Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Graft vs Host Disease; Hematologic Neoplasms; Multiple Myeloma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin

INTERVENTIONS:
Device: Isolex 300i plus MoAbs

SUMMARY:
Cancers of the blood, sometimes referred to as hematologic malignancies, are disorders of bone marrow cells that lead to the failure of the normal function of bone marrow and the uncontrolled growth of cancerous cells in the bone marrow. These cancerous cells can spill over into the bloodstream and affect other organs causing widespread symptoms. The disease is life threatening because it blocks the normal function of the marrow, which is to produce red cells (preventing anemia), white cells (preventing infection), and platelets (preventing progression).

Bone marrow transplants are a potential form of therapy for patients with hematologic malignancies. However, BMT is a complicated procedure and can be associated with dangerous side effects.

In this study researchers are attempting to find ways to reduce the complications of BMT, so that it would be possible to use it more safely and can be offered more patients. In order to do this, researchers are developing new techniques to make BMT safer. It requires making small changes to the standard procedure, which may improve the outcome.

The experimental procedures researchers are evaluating are:

1. <TAB>T-cell depleted peripheral blood progenitor cell (PBPC) transplantation
2. <TAB> Cyclosporine given immediately after the transplant
3. <TAB>Add-back of donor lymphocytes

Patients undergoing these experimental techniques must be monitored closely to see if any benefit or harmful effects will occur. Information gathered from this study can be used to develop further research studies and potential new therapies for hematologic malignancies.

DETAILED DESCRIPTION:
Bone marrow stem cell transplant studies carried out by the NHLBI BMT Unit have focused on approaches to optimize the stem cell and lymphocyte dose in order to improve transplant survival and increase the graft-vs.-leukemia effect. A CD34 stem cell dose of greater than 3 x 10(6)/kg was found to increase survival and reduce relapse, while a CD3+ lymphocyte dose of less than 1 x 10(5)/kg was associated with a very low incidence of GVHD. Although processing of 2 peripheral blood progenitor cell (PBPC) collections with the CellPro immunoabsorption method (combined CD34-positive selection and CD2-negative selection) provided an improvement over previous methods, the system did not always achieve these optimal cell doses. A recent preclinical evaluation by the Department of Transfusion Medicine of a new immunomagnetic cell selection system available from Nexell, Inc. has demonstrated improved recovery of CD34+ cells and increased depletion of T lymphocytes, compared to the CellPro method. Incorporation of the Nexell system (Isolex 300i) into this clinical protocol will allow us to more consistently achieve CD34+ cell doses above the threshold of 3 x 10(6)/kg and CD3+ lymphocyte dosing in the region of 0.5 x 10(5)/kg. This will make it possible to test (1) the potential benefit of optimized transplant cell doses, (2) elimination of post transplant immunosuppression to enhance immune recovery.

In this study, we will use the Nexell Isolex 300i system to obtain more data on the relationship between CD34+ stem cell dose and outcome. In recipients who receive a T cell dose less than 0.5 x 10(5) CD3+ cells/kg the effect of withdrawing cyclosporine on development of GVHD will be evaluated in a cohort study: 20 patients will receive low dose cyclosporine. If the incidence of grade II or worse GVHD is 10% or less, no post transplant immunosuppression will be given to the next cohort and the incidence and severity of acute GVHD again assessed. Stopping rules for unacceptable GVHD severity will be applied. Two match groups HLA 6/6 and 5/6 donor-recipient pairs will be separately studied using this approach.

In a second phase of the study we will continue to accumulate data on T lymphocyte add-back given on day 45 and day 100 after transplant. For this phase, cyclosporine will be reintroduced on day 44 and continued until day 120 to accelerate immune recovery.

Up to 70 patients aged between 10 and 55 years will be studied in each subset (HLA 6/6 and 5/6 matched cohorts). The major endpoint of the study is acute GVHD after transplant. We will also measure engraftment, acute and chronic GVHD, leukemic relapse, transplant-related and all causes of mortality, cytomegalovirus reactivation and leukemia-free survival. Patients will be followed for a minimum of 5 years.

ELIGIBILITY:
* INCLUSION CRITERIA - Patient:

Ages 10-55 years.

Chronic myelogenous leukemia, any of these categories: chronic phase, accelerated phase or blast transformation.

Acute lymphoblastic leukemia, any of these categories: Adults (greater than 18 years) in first remission with high-risk features (presenting leukocyte count greater than 100,000/cu mm, karyotypes t9; 22, t4, t11, biphenotypic leukemia) All second or subsequent remissions, primary induction failure, partially responding or untreated relapse.

Acute myelogenous leukemia (AML): AML in first remission except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), AML t (8;21). All AML in second or subsequent remission, primary induction failure and resistant relapse.

Myelodysplastic syndromes, any of these categories: refractory anemia with transfusion dependence, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia.

Myeloproliferative disorders (myelofibrosis, polycythemia vera, essential thrombocythemia) in transformation to acute leukemia.

Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000 / mcl) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy.

No major organ dysfunction precluding transplantation.

DLCO greater than or equal to 60% predicted.

Left ventricular ejection fraction: greater than or equal to 40% predicted.

ECOG performance status of 0 or 1.

For adults: Written informed consent given by adults. For minors: Written informed consent from one parent or guardian. Informed oral consent from minors: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

Women of childbearing age with a negative pregnancy test may participate.

EXCLUSION CRITERIA - Recipient (any of the following):

Patient pregnant.

Age less than 10 and greater than 55 years.

ECOG performance status of 2 or more.

Severe psychiatric illness in the patient or donor. Mental deficiency sufficiently severe as to make compliance with the treatment unlikely, and making informed consent impossible.

Major anticipated illness or organ failure incompatible with survival from transplant.

DLCO less than 60% predicted.

Left ventricular ejection fraction: less than 40% predicted.

Serum creatinine greater than 3mg/dl.

Serum bilirubin greater than 4 mg/dl.

Transaminases greater than 3x upper limit of normal.

HIV positive (donor or recipient).

History of other malignancies except basal cell or squamous carcinoma of the skin, positive PAP smear and subsequent negative follow up.

Individuals with diseases listed above as eligible for this protocol, but where debility or age makes the risk of intensive myeloablative therapy unacceptable. These patients will be considered for a non-myeloablative allogeneic transplantation protocol (97-H-0202, 99-H-0050).

INCLUSION CRITERIA - Donor:

HLA 6/6 identical or 5/6 (one antigen mismatched) family donor.

Fit to receive G-CSF and give peripheral blood stem cells (normal blood count, normotensive, no history of stroke).

For adults: Written informed consent given by adults. For minors: Written informed consent from one parent or guardian. Informed oral consent from minors: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA - Donor (any of the following):

Pregnant or lactating.

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

HIV positive.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 1999-02-22; Primary Completion 2007-12-28 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with clinically significant acute GHVD (Grade II or higher) following the T depleted PBPC transplant (and before D45 add-back). | Day 45

CONTACTS AND LOCATIONS:
Overall Officials: A. John Barrett, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schmitz N, Dreger P, Suttorp M, Rohwedder EB, Haferlach T, Loffler H, Hunter A, Russell NH. Primary transplantation of allogeneic peripheral blood progenitor cells mobilized by filgrastim (granulocyte colony-stimulating factor). Blood. 1995 Mar 15;85(6):1666-72. PMID 7534141
- [Background] Bensinger WI, Weaver CH, Appelbaum FR, Rowley S, Demirer T, Sanders J, Storb R, Buckner CD. Transplantation of allogeneic peripheral blood stem cells mobilized by recombinant human granulocyte colony-stimulating factor. Blood. 1995 Mar 15;85(6):1655-8. PMID 7534140
- [Background] Veltri S, Smith JW 2nd. Interleukin 1 trials in cancer patients: a review of the toxicity, antitumor and hematopoietic effects. Stem Cells. 1996 Mar;14(2):164-76. doi: 10.1002/stem.140164. PMID 8991536
- [Derived] McIver ZA, Yin F, Hughes T, Battiwalla M, Ito S, Koklanaris E, Haggerty J, Hensel NF, Barrett AJ. Second hematopoietic SCT for leukemia relapsing after myeloablative T cell-depleted transplants does not prolong survival. Bone Marrow Transplant. 2013 Sep;48(9):1192-7. doi: 10.1038/bmt.2013.39. Epub 2013 Mar 25. PMID 23524640
- [Derived] McIver Z, Melenhorst JJ, Wu C, Grim A, Ito S, Cho I, Hensel N, Battiwalla M, Barrett AJ. Donor lymphocyte count and thymic activity predict lymphocyte recovery and outcomes after matched-sibling hematopoietic stem cell transplant. Haematologica. 2013 Mar;98(3):346-52. doi: 10.3324/haematol.2012.072991. Epub 2012 Oct 12. PMID 23065508